CLINICAL TRIAL: NCT07135050
Title: Phase 1/2 First-in-Human Study to Evaluate the Safety, Tolerability, and Efficacy of MZ-1866, an AAV-9 Gene Therapy Delivered by Intracerebroventricular Injection to Participants With Pitt Hopkins Syndrome
Brief Title: Phase 1/2 Study of MZ-1866, an AAV-9 Gene Therapy Delivered by Intracerebroventricular Injection to Participants With Pitt Hopkins Syndrome
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mahzi Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MZ1866-CL101
Record Dates: First submitted 2025-08-04; First posted 2025-08-21 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Pitt Hopkins Syndrome
Keywords: MZ-1866; AAV9 Gene Therapy; Gene Therapy; ICV; Intracerebroventricular; TCF4; PTHS
MeSH Terms: conditions — Pitt-Hopkins syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (MZ-1866) (Experimental): Participants ages 12-25 years
  Interventions: Genetic: MZ-1866
- Cohort 2 (MZ-1866) (Experimental): Participants aged 2-11 years
  Interventions: Genetic: MZ-1866

INTERVENTIONS:
Genetic: MZ-1866 — AAV-9 gene therapy delivered by intracerebroventricular injection

SUMMARY:
The goal of this clinical trial is to learn if MZ-1866 is a safe and tolerable treatment for children and adults with Pitt Hopkins Syndrome.

To evaluate the safety of MZ-1866, the following will be evaluated:

* frequency and severity of adverse events
* physical exam, laboratory results and electrocardiogram findings

Participants will:

* receive a single dose of MZ-1866 by intracerebroventricular injection
* be seen by the study physician and site staff periodically to assess changes to their health status
* be periodically evaluated using neurodevelopmental tools

Caregivers will:

* be interviewed periodically about the health status and development of the participant
* keep diaries and complete periodic questionnaires regarding participant symptoms

ELIGIBILITY:
Inclusion Criteria:

* The participant has a TCF4 gene mutation confirmed as "pathogenic" or "likely pathogenic" by whole exome sequencing, whole genome sequencing, gene panel, single gene testing, or microarray, performed at an accredited laboratory
* Clinical phenotype consistent with Pitt Hopkins Syndrome, in the opinion of the investigator
* The participant, or the participant's parent or legal guardian, is willing to provide access to prior medical records for the collection of demographics and diagnostic and treatment history

Exclusion Criteria:

* A deletion that includes the TCF4 gene that is over 12 Mbp in size
* Another genetic mutation or clinical comorbidity not associated with Pitt Hopkins Syndrome that could potentially confound interpretation of the study data
* A central nervous system structural or vascular abnormality that is a contraindication to the ICV administration procedure, including but not limited to: signs or symptoms of increased intracranial pressure, history of a space-occupying lesion, or presence of a ventricular shunt that would preclude ICV procedures or safety assessments, or increase risk to the participant
* Not able to receive prophylactic corticosteroids due to a medical contraindication or participant has a history of a condition that could worsen with corticosteroid therapy as assessed and determined by the Investigator
* Not able to undergo MRI procedures
* Cannot be anesthetized for the ICV injection

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-03 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of MZ-1866 in participants with Pitt Hopkins Syndrome | Week 104
  Frequency and severity of adverse events of special interest

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of MZ-1866 in participants with Pitt Hopkins Syndrome | Week 104
  Frequency and severity of adverse events
To further assess the safety and tolerability of MZ-1866 in participants with Pitt Hopkins Syndrome | Week 104
  Frequency of clinically significant physical examination findings, vital signs, laboratory tests and electrocardiograms that are considered outside normal range.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Rush University Medical Center, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: Undecided